CLINICAL TRIAL: NCT04967365
Title: Post-Intensive Care Syndrome - Pediatrics (PICS-p): Longitudinal Cohort Study
Acronym: PICS-p
Status: Active, not recruiting | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: Seattle Children's Hospital (Other); Boston Children's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 843844
Record Dates: First submitted 2021-06-28; First posted 2021-07-19 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Critical Illness; Post Intensive Care Unit Syndrome
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case patients: 500 patients who experience greater than or equal to 3 nights in a pediatric ICU with intensive care instrumentation.
- Control patients: 250 patients who experience an overnight stay in a pediatric ICU without intensive care instrumentation.

SUMMARY:
Pediatric Intensive Care Unit (PICU) survival has increased substantially over the past three decades. Currently, an understanding of PICU morbidity and recovery among PICU survivors and their families is limited. Post-intensive care syndrome (PICS) consists of new or worsening impairments in physical, cognitive, or mental health status that arise and may persist after critical illness. The characteristics of PICS in children (PICS-p) are unknown. The objective of this study is to learn about pediatric recovery from critical illness to guide future intervention research to optimize child and family health.

DETAILED DESCRIPTION:
PICS-p is a prospective longitudinal cohort study of pediatric patients experiencing 3 or more days of intensive care therapies at one of approximately 30 U.S. PICUs to evaluate child and family outcomes over two years post-PICU discharge. We will compare outcomes of these PICU patients with a control group of patients who received an overnight PICU stay but did not receive intensive care therapies, as well as with published quality of life data from the general and chronically ill populations. Children and their families will be enrolled locally from each PICU, their baseline data will be collected by local research staff, and their post-discharge outcomes will be followed centrally from the University of Pennsylvania and the Seattle Children's Research Institute. Our specific aims are to determine the physical, cognitive, emotional, and social health outcomes and trajectory of recovery in a population of children post-critical illness; to determine the baseline health, presenting problem, and PICU factors associated with impaired physical, cognitive, emotional, and social outcomes among PICU survivors; and to determine the emotional and social health outcomes in parents and siblings of PICU survivors. Our primary goal is to explicate the impact of pediatric critical illness over a two-year period of time to guide future intervention research to optimize child and family outcomes. Our overall goal is to improve the health and well-being of PICU survivors and their families.

ELIGIBILITY:
Case Inclusion criteria:

1. Current admission is the child's first PICU (including pediatric subspecialty ICU) admission
2. Patient age ≥4 weeks and ≥44 weeks corrected gestational age and <16 years (has not yet reached 16th birthday) on PICU admission
3. At least one parent/legal guardian (≥18 years of age or considered emancipated) living with the potential subject
4. PICU LOS of 3 days (covering at least 3 nights from midnight to 7am) in which the patient received intensive care therapies for organ dysfunction (for example, invasive mechanical ventilation, vasopressors/inotropes, acute renal replacement therapy, or other extracorporeal therapies).
5. Anticipated patient discharge to home (directly or indirectly after a stay in another facility)

Case Exclusion criteria:

1. Patient history of neonatal intensive care unit hospitalization
2. Life expectancy not anticipated to be more than one year (e.g., active do not resuscitate [DNR] plan or actively managed by the palliative care team for end-of-life symptom management)
3. Patient in foster care or ward of the state

Control subjects: As above but will be PICU patients who received an overnight PICU stay (<36 hours covering one midnight to 7am time period) that did not include intensive care therapies. Post-operative children who were intubated/extubated in the operating room/PACU (or intubated in the operating room and extubated in the PICU on arrival and prior to parent presence at the bedside) can be enrolled as control subjects. Control subjects will be frequency matched to cases on age group, sex, and medical complexity, that is, complex chronic disease (C-CD), noncomplex chronic disease (NC-CD), and without CD on a 2:1 case:control ratio.

Family Subjects: At least one eligible parent/legal guardian must be willing to participate. In addition, up to two cognitively capable siblings (PCPC of 1 or 2) aged 8 to <16 years, who live with the patient, and who have not been ICU hospitalized will be invited to participate. If more than two siblings are eligible, the two siblings with the next birthday (regardless of birth year) will be invited to participate.

Ages: 1 Month to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patents surviving a pediatric intensive care unit hospitalization
Sampling Method: Probability Sample
Enrollment: 755 (Actual)
Dates: Start 2021-07-27 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Health related quality of life (HRQOL) - Patient | Two years
  PedsQL™ 4.0 Generic Core or Infant Scales (self report)
Health related quality of life (HRQOL) - Parent | Two years
  PedsQL™ 4.0 Generic Core or Infant Scales (parent report)

SECONDARY OUTCOMES:
Fatigue - Patient | Two Years
  PedsQL™ Multidimensional Fatigue Scale v3.0 (self report)
Fatigue - Parent | Two Years
  PedsQL™ Multidimensional Fatigue Scale v3.0 (parent report)
Sleep - Patient | Two Years
  PROMIS Pediatric Sleep Disturbance - Short Form 4a and Pediatric Sleep-Related Impairment - Short Form 4a (self report)
Sleep - Parent | Two Years
  PROMIS Sleep Disturbance - Short Form 4a and Sleep-Related Impairment - Short Form 4a (parent report)
Cognitive Functioning - Patient | Two Years
  PedsQL™ Cognitive Functioning Scale and Pediatric Cerebral Performance Category (PCPC)
Cognitive Functioning - Parent | Two Years
  PedsQL™ Cognitive Functioning Scale (parent report) and Pediatric Cerebral Performance Category (PCPC) (parent report)
Pain - Patient | Two Years
  PedsQL™ Pediatric Pain Questionnaire and PROMIS Pediatric Pain Interference - Short Form 8a (self report)
Post Traumatic Stress Disorder (PTSD)- Patient | Two Years
  Child PTSD Symptom Scale for DSM-5 (CPSS-V) (self report)
Post Traumatic Stress Disorder (PTSD)- Parent | Two Years
  Young Child PTSD Screen - Revised PICU (YCPS R - PICU) (parent report); PTSD Checklist for DSM-5 (PCL-5) (parent report)
Strengths and Difficulties - Patient | Two Years
  Strengths and Difficulties Questionnaire (SDQ)
Strengths and Difficulties - Sibling | Two Years
  Strengths and Difficulties Questionnaire (SDQ)
Hope - Patient | Two Years
  Children's Hope Scale (CHS)
Hope - Sibling | Two Years
  Children's Hope Scale (CHS)
Growth and Development - Patient | Two Years
  Survey of Well-being of Young Children (SWYC) - Milestones only (parent report)
Functional status - Patient | Two Years
  Functional Status Scale (FSS) and Pediatric Overall Performance Category (POPC) (parent report)
Family impact | Two years
  PedsQL™ Family Impact Module v2.0 (parent report)
Growth - Parent | Two Years
  Post-traumatic Growth Inventory - Short Form (PTGI-SF) (parent self report)
Depression - Parent | Two years
  Patient Health Questionnaire-4 (PHQ-4) (parent self report)
HRQOL - Sibling | Two Years
  PedsQL Version 4.0 Generic Core Scales (sibling self report)
Caregiving - Sibling | Two Years
  Multidimensional Assessment of Caring Activities (MACA-YC18) (sibling self report)

CONTACTS AND LOCATIONS:
Overall Officials: Martha AQ Curley, RN, PhD, Principal Investigator — University of Pennsylvania; R. Scott Watson, MD, Principal Investigator — Seattle Children's Hospital
Locations (30):
- United States (30):
  - Alabama Children's Hospital, Birmingham, Alabama
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Annopinder Bhalla MD, Los Angeles, California
  - Lucille Packard Children's Hospital Stanford, Palo Alto, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's National Hospital, Washington D.C., District of Columbia
  - Children's Hospital of Atlanta, Atlanta, Georgia
  - Ann & Robert H Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Comer Children's Hospital, Chicago, Illinois
  - Riley Children's Health at Indiana University, Indianapolis, Indiana
  - Norton Children's Hospital, Louisville, Kentucky
  - Charlotte R Bloomberg Children's Center, Baltimore, Maryland
  - CS Mott Children's Hospital, Detroit, Michigan
  - Massonic Children's Hospital, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - St Louis Children's Hospital, St Louis, Missouri
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - UNC Children's Hospital Chapel Hill, Chapel Hill, North Carolina
  - Brenner Children's Hospital, Winston-Salem, North Carolina
  - Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Doernbecher Children's Hospital, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - LeBonheur Children's Hospital, Memphis, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Children's Medical Center Dallas, Dallas, Texas
  - Texas Children's Hospital, Houston, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - Children's Hospital of Richmond, Richmond, Virginia
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Curley MAQ, Watson RS, Killien EY, Kalvas LB, Perry-Eaddy MA, Cassidy AM, Miller EB, Talukder M, Manning JC, Pinto NP, Rennick JE, Colville G, Asaro LA, Wypij D. Design and rationale of the Post-Intensive Care Syndrome - paediatrics (PICS-p) Longitudinal Cohort Study. BMJ Open. 2024 Feb 24;14(2):e084445. doi: 10.1136/bmjopen-2024-084445. PMID 38401903